CLINICAL TRIAL: NCT02170519
Title: Inhaled Aerosolized Prostacyclin for Pulmonary Hypertension Requiring Inhaled Nitric Oxide
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Project was completed
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013737
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2014-06

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 2: Inhaled Iloprost continuous (Experimental): Each subject will have a stable dose of INO therapy as established by the attending physicians for at least one hour. Initial baseline data collection will then be made.
  A 20 mcg dose of Iloprost will be given initially. During this treatment there will be a nitric oxide titration to 0. Iloprost will be aerosolized continuously at a dose of 5-30mcg/hour for as long as the attending physician deems it necessary to deliver vasodilator therapy.
  Interventions: Drug: Inhaled Iloprost
- Phase 1: Inhaled Iloprost 3 doses (Experimental): Each subject will have a stable dose of INO therapy as established by the attending physicians for at least one hour. Initial baseline data collection will then be made.
  A 20 mcg dose of Iloprost will be given initially. During this treatment there will be a nitric oxide titration to 0. Iloprost will be aerosolized three different times on hour apart. Thirty minutes after the last iloprost dose, INO will be added back at the previous (baseline) dose.
  Interventions: Drug: Inhaled Iloprost

INTERVENTIONS:
Drug: Inhaled Iloprost — A 20 mcg dose of Iloprost will be given initially.
  Other Names: Ventavis

SUMMARY:
Acute secondary pulmonary hypertension (PH) often leads to dysfunction of the right ventricle (RV) and can be a significant cause of patient morbidity and mortality. Selective pulmonary vasodilation with inhaled nitric oxide (INO) has become the treatment of choice for this condition. The evidence supporting INO safety and efficacy under these circumstances is sparse, however, and is largely extrapolated from the use of INO in neonatal pulmonary hypertension. Moreover, the high cost and potential toxicity of INO makes the therapy far from ideal. Emerging evidence suggests that inhaled aerosolized prostacyclins such as iloprost may be a favorable alternative therapy.

DETAILED DESCRIPTION:
Phase 1- In the original study, 3 doses of Iloprost were given. This was revised after 5 subjects were enrolled in order to study the effects of continuous delivery over a longer period of time.

Phase 2 - All remaining subjects received Iloprost as a continuous treatment.

The study was designed for an enrollment of 200 subjects and was ended early.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical evidence of pulmonary hypertension (PH) requiring INO therapy as prescribed by the attending physician.
2. Indwelling arterial catheter.
3. Signed informed consent

Exclusion Criteria:

1. Clinically unstable circulatory condition requiring epinephrine > 0.1 mcg/kg/min or levophed, or already meeting treatment failure criteria (see section 5.3 below)
2. Known hypersensitivity to prostacyclin compounds
3. Patients receiving sildenafil or bosentan
4. Refusal by the attending physician

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil MacIntyre, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2: Inhaled Iloprost Continuous: Each subject will have a stable dose of INO therapy as established by the attending physicians for at least one hour. Initial baseline data collection will then be made.
  A 20 mcg dose of Iloprost will be given initially. During this treatment there will be a nitric oxide titration to 0. Iloprost will be aerosolized continuously at a dose of 5-30mcg/hour for as long as the attending physician deems it necessary to deliver vasodilator therapy.
  Inhaled Iloprost: A 20 mcg dose of Iloprost will be given initially.
- Phase 1: Inhaled Iloprost 3 Doses: Each subject will have a stable dose of INO therapy as established by the attending physicians for at least one hour. Initial baseline data collection will then be made.
  A 20 mcg dose of Iloprost will be given initially. During this treatment there will be a nitric oxide titration to 0. Iloprost will be aerosolized three different times on hour apart. Thirty minutes after the last iloprost dose, INO will be added back at the previous (baseline) dose.
  Inhaled Iloprost: A 20 mcg dose of Iloprost will be given initially.
Period: Overall Study
Arm/Group | Phase 2: Inhaled Iloprost Continuous | Phase 1: Inhaled Iloprost 3 Doses
Started | 22 | 5
Completed | 22 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 2: Inhaled Iloprost Continuous | Phase 1: Inhaled Iloprost 3 Doses | Total
Number analyzed (Participants) | 22 | 5 | 27
Age, Customized [Number; unit: participants]
  >18 years | 21 | 5 | 26
  <=18 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 1 | 15
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 22 | 5 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Oxygen Saturation (SpO2) From Baseline
Description: Readings were taken from the medical record and the data may not have been present at the exact time frames.
Time Frame: 30 mins after initial dose, every 2 hours as long as subject was on drug up to approximately 24 hours
Population: Phase 2 subjects
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 2: Inhaled Iloprost Continuous
Number analyzed (Participants) | 22
percent change
  30 mins after initial dose | -0.4 (1.7)
  2 hours | -0.8 (2.8)
  4 hours | -1.2 (2.9)
  6 hours | -0.2 (3.6)
  8 hours | -0.7 (3.1)
  10 hours | -0.9 (3.0)
  12 hours | -0.9 (3.7)
  18 hours | -1.5 (5.6)
  24 hours | 1.7 (6.4)

2. Primary Outcome: Percent Change in Oxygen Saturation (SpO2) From Baseline
Time Frame: dose 1 (1 hour), dose 2 (2 hour), dose 3 (3 hour), combined therapy (4.5 - 5 hour), end INO (6 - 7 hour)
Population: Phase 1 subjects
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Phase 1: Inhaled Iloprost 3 Doses: Each subject will have a stable dose of INO therapy as established by the attending physicians for at least one hour. Initial baseline data collection will then be made.
  A 20 mcg dose of Iloprost will be given initially. During this treatment there will be a nitric oxide titration to 0. Iloprost will be aerosolized three different times on hour apart. Thirty minutes after the last iloprost dose, INO will be added back at the previous (baseline) dose and data collected 5 minutes later (combined therapy). Another 1 hour period of stable baseline dose INO therapy will be given during which the final data collection will occur (end INO).
  Inhaled Iloprost: A 20 mcg dose of Iloprost will be given initially.
Arm/Group | Phase 1: Inhaled Iloprost 3 Doses
Number analyzed (Participants) | 5
percent change
  dose 1 | -0.4 (0.6)
  dose 2 | -0.4 (1.6)
  dose 3 | 0.0 (2.9)
  combined therapy | 0.2 (2.4)
  end INO | 0.4 (1.6)

3. Primary Outcome: Change in Mean Heart Rate From Baseline
Time Frame: 30 mins after initial dose, every 2 hours as long as subject was on drug up to approximately 24 hours
Population: Phase 2 subjects
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 2: Inhaled Iloprost Continuous
Number analyzed (Participants) | 22
percent change
  30 mins after initial dose | -1.8 (4.4)
  2 hours | -1.1 (6.6)
  4 hours | 4.2 (18.7)
  6 hours | 0.8 (12.5)
  8 hours | -1.0 (13.7)
  10 hours | 2.2 (14.3)
  12 hours | -2.9 (12.0)
  18 hours | -4.0 (12.6)
  24 hours | -9.9 (16.1)

4. Primary Outcome: Change in Mean Heart Rate From Baseline
Time Frame: dose 1 (1 hour), dose 2 (2 hour), dose 3 (3 hour), combined therapy (4.5 - 5 hour), end INO (6 - 7 hour)
Population: Phase 1 subjects
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 1: Inhaled Iloprost 3 Doses
Number analyzed (Participants) | 5
percent change
  dose 1 | 0.9 (4.8)
  dose 2 | 2.5 (4.5)
  dose 3 | 0.7 (6.7)
  combined therapy | 0.9 (7.8)
  end INO | -0.2 (8.9)

5. Secondary Outcome: Change in Cardiac Output (CO) From Baseline
Time Frame: 30 mins after initial dose, every 2 hours as long as subject was on drug up to approximately 24 hours
Population: Phase 2 subjects: 4 subjects did not have a swan ganz catheter. 1 subject had a swan ganz catheter, but measurement was unattainable.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 2: Inhaled Iloprost Continuous
Number analyzed (Participants) | 17
percent change
  30 mins after initial dose | 16.2 (25.6)
  2 hours | 3.4 (20.5)
  4 hours | 21.2 (31.1)
  6 hours | 14.3 (43.1)
  8 hours | 12.5 (55.1)
  10 hours | 9.3 (43.3)
  12 hours | 8.9 (38.8)
  18 hours | 36.6 (68.9)
  24 hours | 4.4 (27.9)

6. Secondary Outcome: Change in Cardiac Output (CO) From Baseline
Time Frame: dose 1 (1 hour), dose 2 (2 hour), dose 3 (3 hour), combined therapy (4.5 - 5 hour), end INO (6 - 7 hour)
Population: Phase 1 subjects
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 1: Inhaled Iloprost 3 Doses
Number analyzed (Participants) | 5
percent change
  dose 1 | 8.4 (33.7)
  dose 2 | -0.9 (36.3)
  dose 3 | 8.7 (18.6)
  combined therapy | 2.5 (9.3)
  end INO | -8.7 (20.9)

7. Primary Outcome: Number of Treatment Failures
Description: Treatment failure is defined as Central venous pressure (CVP) ≥ 20 mm Hg and any one of the following:
  1. Cardiac Index (CI) >/= 1.8 L/min/m2
  2. Administration of >/=0.1 ug/kg/min Epinephrine or Norepinephrine
  3. MAP </= 50 mmHg (or as appropriate for age in pediatrics).
  4. SvO2</= 55% (or < 45% for patients with R to L intracardiac shunting and, thus, cyanosis at baseline.}
Time Frame: as long as subject was on drug up to approximately 24 hours
Measure: Number; unit: participants
Arm/Group | Phase 2: Inhaled Iloprost Continuous | Phase 1: Inhaled Iloprost 3 Doses
Number analyzed (Participants) | 22 | 5
participants | 0 | 0

8. Primary Outcome: Change in Mean Pulmonary Artery Pressure (mPAP) From Baseline
Time Frame: 30 mins after initial dose, every 2 hours as long as subject was on drug up to approximately 24 hours
Population: Phase 2 subjects: Measurement completed on subjects having a Swan Ganz catheter. 4 subjects did not have a swan ganz catheter.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 2: Inhaled Iloprost Continuous
Number analyzed (Participants) | 18
percent change
  30 mins after initial dose | 1.9 (9.6)
  2 hours | -1.1 (19.1)
  4 hours | 3.1 (17.2)
  6 hours | -1.9 (16.9)
  8 hours | -3.2 (20.4)
  10 hours | 1.6 (12.7)
  12 hours | 1.3 (15.7)
  18 hours | 6.5 (17.1)
  24 hours | 7.0 (23.5)

9. Primary Outcome: Change in Mean Pulmonary Artery Pressure (mPAP) From Baseline
Time Frame: dose 1 (1 hour), dose 2 (2 hour), dose 3 (3 hour), combined therapy (4.5 - 5 hour), end INO (6 - 7 hour)
Population: Phase 1 subjects
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 1: Inhaled Iloprost 3 Doses
Number analyzed (Participants) | 5
percent change
  dose 1 | -0.9 (10)
  dose 2 | -6.5 (10.9)
  dose 3 | -10.2 (8.6)
  combined therapy | -13.0 (9.6)
  end INO | -9.3 (12.9)

10. Secondary Outcome: Change in Mean Venous Oxygen Saturation (SvO2) From Baseline
Description: SvO2 represents an average of all the venous oxygen saturations of the various organs and tissues.
Time Frame: 30 mins after initial dose, every 2 hours as long as subject was on drug up to approximately 24 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 2: Inhaled Iloprost Continuous
Number analyzed (Participants) | 17
percent change
  30 mins after initial dose | 1.5 (8.5)
  2 hours | 1.5 (9.6)
  4 hours | 1.3 (5.1)
  6 hours | 1.1 (7.4)
  8 hours | 1.4 (4.8)
  10 hours | -3.4 (7.4)
  12 hours | -1.6 (6.6)
  18 hours | -0.5 (10.3)
  24 hours | -3.0 (13.9)

11. Secondary Outcome: Change in Mean Venous Oxygen Saturation (SvO2) From Baseline
Time Frame: dose 1 (1 hour), dose 2 (2 hour), dose 3 (3 hour), combined therapy (4.5 - 5 hour), end INO (6 - 7 hour)
Population: Phase 1 subjects
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 1: Inhaled Iloprost 3 Doses
Number analyzed (Participants) | 5
percent change
  dose 1 | -2.3 (2.3)
  dose 2 | -2.6 (5.5)
  dose 3 | -1.7 (7.5)
  combined therapy | 0.3 (6.0)
  end INO | 1.4 (2.0)

ADVERSE EVENTS:
Arm/Group | Phase 2: Inhaled Iloprost Continuous | Phase 1: Inhaled Iloprost 3 Doses
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/5
Other Adverse Events (participants affected / at risk) | 0/22 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes